CLINICAL TRIAL: NCT05819398
Title: Randomised, Double-blind, Placebo-controlled, Phase IIb/Phase III Study to Evaluate the Efficacy and Safety of Spesolimab in Patients With Moderate to Severe Hidradenitis Suppurativa. Lunsayil 1.
Brief Title: Lunsayil 1: A Study to Test Whether Spesolimab Helps People With a Skin Disease Called Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0098; 2022-501074-19-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Spesolimab low dose group (Experimental): Patients with moderate to severe HS were administered an initial weekly low dose of spesolimab via i.v. (Week 0 to Week 3). Afterwards, patients were administered a lower weekly s.c. dose of spesolimab for 4 weeks (Week 4 to Week 7). Patients were then administered a maintenance s.c. dose of spesolimab every two weeks until the end of the treatment (Week 8 to Week 48).
  From Week 16, if patients had inadequate clinical response defined as 25% increase in the ANdT count compared to baseline, the dose could be increased every two weeks to a pre-determined concentration.
  Interventions: Drug: Spesolimab i.v.; Drug: Spesolimab s.c.
- Spesolimab medium dose group (Experimental): Patients with moderate to severe HS were administered an initial weekly medium dose of spesolimab via i.v. (Week 0 to Week 3). Afterwards, patients were administered a lower weekly s.c. dose of spesolimab for 4 weeks (Week 4 to Week 7). Patients were then administered a maintenance s.c. dose of spesolimab every two weeks until the end of the treatment (Week 8 to Week 48).
  Interventions: Drug: Spesolimab i.v.; Drug: Spesolimab s.c.
- Spesolimab high dose group (Experimental): Patients with moderate to severe HS were administered an initial weekly high dose of spesolimab via i.v. (Week 0 to Week 3). Afterwards, patients were administered a lower weekly s.c. dose of spesolimab for 4 weeks (Week 4 to Week 7). Patients were then administered a maintenance s.c. dose of spesolimab every two weeks until the end of the treatment (Week 8 to Week 48).
  Interventions: Drug: Spesolimab i.v.; Drug: Spesolimab s.c.
- Placebo (Placebo Comparator): Patients with moderate to severe Hidradenitis suppurativa (HS) were administered an initial weekly dose of placebo via intravenous infusion (i.v.) (Week 0 to Week 3). Afterwards, patients were administered a subcutaneous injection (s.c.) dose of placebo once a week for 4 weeks (Week 4 to Week 7), and once every 2 weeks for the following 7 weeks (Week 8 to Week 14).
  From Week 16 until the end of treatment (Week 48), patients were switched to the same s.c. dose of spesolimab administered to patients in the medium and high dose groups (starting with 3 loading s.c. doses of spesolimab every week and then maintenance s.c. dose of spesolimab every 2 weeks).
  Interventions: Drug: Spesolimab s.c.; Drug: Placebo matching Spesolimab i.v.; Drug: Placebo matching Spesolimab s.c.

INTERVENTIONS:
Drug: Spesolimab i.v. — Weekly dose of spesolimab via i.v. for 4 weeks.
  Other Names: Spevigo®
  Arms: Spesolimab high dose group; Spesolimab low dose group; Spesolimab medium dose group
Drug: Spesolimab s.c. — Weekly s.c. dose of spesolimab for 4 weeks (3 weeks for Placebo), and maintenance s.c. dose of spesolimab every two weeks until the end of the treatment.
  Other Names: Spevigo®
Drug: Placebo matching Spesolimab i.v. — Weekly dose of placebo via i.v. for 4 weeks.
  Arms: Placebo
Drug: Placebo matching Spesolimab s.c. — Weekly s.c. dose of placebo for 4 weeks, and once every 2 weeks for the following 7 weeks.
  Arms: Placebo

SUMMARY:
This study is open to adults with moderate to severe hidradenitis suppurativa (HS). The purpose of this study is to find out whether a medicine called spesolimab helps people with HS. People who have previously taken specific medicines such as immunosuppressive biologics other than Tumor necrosis factor (TNF) inhibitors cannot take part.

This study has 2 parts. In Part 1, participants are divided into 4 groups of almost equal size. 3 groups get different doses of spesolimab, 1 group gets placebo. All participants get injections into a vein or under the skin. Placebo injections look like spesolimab injections, but do not contain any medicine. Every participant has an equal chance of being in each group. In the beginning, participants get the study medicine every week and later every 2 weeks. After 4 months, participants in the placebo group switch to spesolimab treatment.

In Part 2, participants are divided into 2 groups. One group gets a suitable dose of spesolimab that was found in Part 1 of the study. The other group gets placebo. After 4 months, participants in the placebo group switch to spesolimab treatment.

Participants join only one of the two parts. They are in the study for about 1 year. During this time, they visit the study site in the beginning every week and later every 2 weeks. Some of the visits can be done at the participant's home instead of the study site. The doctors regularly check participants' HS symptoms. The results are compared between the groups to see whether spesolimab works. The doctors also regularly check participants' general health and take note of any unwanted effects.

DETAILED DESCRIPTION:
Main endpoints for Part 2 will be supported by Part 1 results available at time of primary analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Of full age of consent at screening.
2. Signed and dated written informed consent in accordance with International Council on Harmonisation-Good clinical practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Moderate to severe HS.
4. HS lesions in at least 2 distinct anatomic areas.
5. Biologic naive or Tumor Necrosis Factor inhibitor (TNFi)-exposed for HS.
6. For biologic naïve, inadequate response to an adequate course of appropriate oral antibiotics for treatment of HS in the last 1 year prior to the Baseline visit, as per investigator discretion. All participants must have previous exposure to antibiotics for HS.
7. Total AN count of greater than or equal to 5.
8. Total dT count of at least 1 at Baseline visit. Further inclusion criteria apply.

Exclusion Criteria:

1. Participants who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
2. Prior exposure to any immunosuppressive/immunomodulatory biologic other than TNFi for HS.
3. Prior exposure to Interleukin 36 receptor (IL-36R) inhibitors including spesolimab.
4. Treated with any investigational device or investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives of the drug, whichever is longer.
5. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
6. Participants with history of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients.
7. Participants with a transplanted organ (with exception of a corneal transplant >12 weeks prior to screening) or who has ever received stem cell therapy (e.g., Remestemcel-L).
8. Participants with any documented active or suspected malignancy or history of malignancy within 5 years prior to the screening visit, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ carcinoma of uterine cervix.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (162):
- United States (19):
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Integrative Skin Science and Research-Sacramento-69402, Sacramento, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Ziaderm Research, North Miami Beach, Florida
  - ForCare Clinical Research, Inc., Tampa, Florida
  - Olympian Clinical Research-Tampa-69560, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC-Indianapolis -68995, Indianapolis, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Oakland Hills Dermatology, PC, Auburn Hills, Michigan
  - Skin Specialists, P.C., Omaha, Nebraska
  - AXIS Clinicals, Fargo, North Dakota
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Clinical Trial Services, Greenville, South Carolina
  - Center for Clinical Studies-Houston-58806, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Argentina (6):
  - STAT Research, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Hospital Alemán, Capital Federal
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Instituto de Especialidades de la Salud Rosario, Rosario
  - Sanatorio 9 de Julio S.A., San Miguel de Tucumán
- Australia (3):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Alfred Hospital, Melbourne, Victoria
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire de Liège, Liège
- Bulgaria (6):
  - Medical Center "Kordis", Pleven
  - ASMC-IPSMC-skin and Veneral Diseases, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - DCC "Fokus-5-LZIP" OOD, Sofia
  - Medical Military Academy MHAT Sofia, Sofia
  - MHAT Prof Stoyan Kirkovich AD, Stara Zagora
- Canada (5):
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
- Chile (2):
  - Centro Internacional de Estudios Clínicos (CIEC), Comuna de Recoleta
  - Clínica Dermacross S.A., Vitacura
- China (9):
  - Peking University First Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Southern Medical University Dermatology Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Shanghai Skin Disease Hospital, Shanghai
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi
  - Wuhan Union Hospital, Wuhan
- Czechia (4):
  - University Hospital Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, Plzen-Bory
  - Univ. Hospital Kralovske Vinohrady, Prague
  - University Hospital Bulovka, Prague
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg og Frederiksberg Hospital, København NV
  - Sjællands Universitetshospital, Roskilde
- Suomen Terveystalo oy Tampere, Tampere, Finland
- France (7):
  - HOP Privé Antony, Antony
  - HOP Edouard Herriot, Lyon
  - HOP Timone, Marseille
  - HOP l'Archet, Nice
  - HOP Saint-Louis, Paris
  - HOP la Milétrie, Poitiers
  - HOP Pontchaillou, Rennes
- Germany (6):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite Universitätsmedizin Berlin KöR, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Hautmedizin Saar, Merzig
  - Klinikum Oldenburg AöR, Oldenburg
- Greece (5):
  - University General Hospital Attikon, Athens
  - Attikon University Hospital, Athens
  - Andreas Syggros Hospital of Cutaneous & Venereal Diseases, Athens
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
- Israel (5):
  - Haemek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sheba MC, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Pol. Universitario Tor Vergata, Roma
  - Istituto Dermopatico Dell'Immacolata - IDI - IRCCS, Roma
- Japan (18):
  - Japan Community Healthcare Organization Chukyo Hospital, Aichi, Nagoya
  - Nagoya City University Hospital, Aichi, Nagoya
  - Fujita Health University Hospital, Aichi, Toyoake
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Fukuoka, Kurume
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Meiwa Hospital, Hyogo, Nishinomiya
  - University of Tsukuba Hospital, Ibaraki, Tsukuba
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama
  - University of the Ryukyus Hospital, Okinawa, Ginowan
  - Kansai Medical University Hospital, Osaka, Hirakata
  - Shiga University of Medical Science Hospital, Shiga, Otsu
  - Dokkyo Medical University Hospital, Tochigi, Shimotsuga-gun
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital, Santariskiu, Vilnius
- Malaysia (8):
  - Hospital Pulau Pinang-Pulau Pinang-21953, Georgetown Pulau Pinang
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu
  - Sarawak General Hospital, Kuching
  - Sunway Medical Centre, Selangor Darul Ehsan
- Mexico (5):
  - Derma Norte del Bajio S.C., Aguascalientes
  - Grupo Clinico CATEI S.C., Guadalajara
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Eukarya Pharmasite, Monterrey
  - Arke SMO S.A. de C.V., Veracruz
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Waikato Hospital, Hamilton, New Zealand
- Philippines (4):
  - Southern Philippines Medical Center -Davao-62091, Davao City
  - Center for Skin Research, Testing and Product Development, Makati City
  - Philippine General Hospital, Manila, Philippines
  - East Avenue Medical Center, Quezon City
- Poland (8):
  - Non-Public Health Care Facility LABDERM, Ossy
  - NSZOZ Termedica Clinical Research Center, Poznan
  - Frederic Chopin University Hospital No. 1 in Rzeszow, Rzeszów
  - High-Med Specialist Clinic, Warsaw, Warsaw
  - National Medical Institute MSWiA, Warsaw
  - Provita Clinic, Warsaw
  - Royalderm, Warsaw
  - Centrum Zdrowia WroMedica, Wroclaw
- National University Hospital-Singapore-42005, Singapore, Singapore
- Slovakia (2):
  - DOST sro - Sanatorium-Type Dermatovenereological Department, Svidník
  - FN Trnava, Trnava
- TASK Applied Science, Cape Town, South Africa
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (10):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía-Córdoba-40500, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital General de Granollers, Granollers
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Manises, Manises
  - Hospital Universitario de Salamanca, Salamanca
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Miguel Servet, Zaragoza
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - University Hospital Bern/Inselspital Bern, Bern
  - Hôpitaux Universitaires Genève (HUG), Geneva
- Chang Gung Memorial Hospital Linkou, Taoyuan District, Taiwan
- Turkey (Türkiye) (3):
  - SBU Gulhane Training and Research Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
- United Kingdom (2):
  - Gloucestershire Royal Hospital, Gloucester
  - St George's Hospital-London-26733, London
- HCMC Hospital of Dermato-Venereology-Ho Chi Minh-66092, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an international, Phase IIb/III multi-center, double-blind, placebo-controlled, randomised trial assessing the efficacy and safety of spesolimab versus placebo in patients with moderate to severe Hidradenitis suppurativa.
Pre-assignment Details: Subjects were screened for eligibility prior to participation and attended a specialist site which ensured that they met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. The trial was completed according to the protocol. However, part 2 was never initiated. The primary and interim analyses of part 1 (dose finding phase) didn't show signal to proceed with the confirmatory phase (part 2).
Period: Overall Study
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Started | 53 | 53 | 52 | 51
Completed | 21 | 20 | 20 | 17
Not Completed | 32 | 33 | 32 | 34
Not completed — Withdrawal by Subject | 11 | 7 | 6 | 6
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1
Not completed — Adverse Event | 1 | 3 | 4 | 5
Not completed — Other than listed | 0 | 2 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 20 | 18 | 20 | 22

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group | Total
Number analyzed (Participants) | 53 | 53 | 52 | 51 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (8.8) | 37.0 (12.1) | 39.5 (13.9) | 39.2 (13.5) | 37.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 20 | 20 | 81
  Male | 34 | 31 | 32 | 31 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 7 | 27
  Not Hispanic or Latino | 42 | 44 | 44 | 42 | 172
  Unknown or Not Reported | 5 | 2 | 1 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 2 | 5
  Asian | 22 | 13 | 13 | 15 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 3 | 9
  White | 23 | 34 | 35 | 29 | 121
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 5 | 2 | 1 | 2 | 10
Number of draining fistulas/tunnels (dT) [Mean (Standard Deviation); unit: Draining fistulas/tunnels] — Tunnel/fistula/sinus should be counted as dT only if draining. Baseline values were recorded prior to first drug administration at Week 0.
  Draining fistulas/tunnels | 5.2 (5.8) | 5.1 (5.1) | 7.0 (10.9) | 6.5 (6.7) | 5.9 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Percent Change From Baseline in Draining Fistula/Tunnel (dT) Count at Week 8
Description: Percent change from baseline in draining fistula/tunnel (dT) count at Week 8 is reported. Tunnel/fistula/sinus were counted as dT only if draining. Percent change was calculated as follows: (dT count at week 8 - dT count at baseline)/ dT at baseline.
  Least square means and standard errors were estimated by Mixed effect model for repeated measurements (MMRM). The MMRM included fixed categorical effects of treatment at each visit, Tumor Necrosis Factor inhibitor (TNFi) status at baseline, and categorical baseline dT count at each visit. Visit were treated as the repeated measure with an unstructured covariance structure used to model the within-trial participant measurements.
Time Frame: The MMRM model incorporates dT count from baseline (Week 0), Week 2, Week 4, Week 6 and Week 8. The data represent the Least Squares Means at Week 8.
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug. The use of "treatment policy" approach disregards the intercurrent event and uses the value of the variable regardless of the occurrence of the intercurrent event.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Number analyzed (Participants) | 53 | 53 | 52 | 51
Percentage change | -21.5 (7.7) | -41.9 (7.8) | -39.3 (7.9) | -25.8 (7.9)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab low dose group; The MMRM included fixed categorical effects of treatment at each visit, Tumor Necrosis Factor inhibitor (TNFi) status at baseline, and categorical baseline dT count at each visit. Visit were treated as the repeated measure with an unstructured covariance structure used to model the within-trial participant measurements; Test type: Other; Difference of least square means = -20.4, 95% CI 2-sided [-41.9 to 1.1], Standard Error of Mean 10.9 — Difference = (least square mean Spesolimab low dose) - (least square mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs Spesolimab medium dose group; [analysis description as in outcome 1, analysis 1]; Test type: Other; Difference of least square means = -17.8, 95% CI 2-sided [-39.5 to 3.9], Standard Error of Mean 11.0 — Difference = (least square mean Spesolimab medium dose) - (least square mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 1]; Test type: Other; Difference of least square means = -4.3, 95% CI 2-sided [-26.0 to 17.5], Standard Error of Mean 11.0 — Difference = (least square mean Spesolimab high dose) - (least square mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; Multiple comparison and modelling techniques (MCPMod) was used to evaluate several possible dose response models (patterns: Linear, Exponential, Emax, SigEmax, BetaMod), and to identify the best-fitting model or subset of models; Test type: Other; p = 0.697, MCPMod Linear model — Adjusted p-value from multiple contrast test; No assumptions
Statistical Analysis 5: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.844, MCPMod Exponential: model — Adjusted p-value from multiple contrast test; Assumption: 30% of the maximum effect is achieved at the medium dose
Statistical Analysis 6: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.256, MCPMod Emax model — Adjusted p-value from multiple contrast test; Assumption: 70% of the maximum effect is achieved at the medium dose
Statistical Analysis 7: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.571, MCPMod SigEmax model — Adjusted p-value from multiple contrast test; Assumption: 70% of the maximum effect is achieved at the medium dose and 25% of the maximum effect is achieved at the low dose
Statistical Analysis 8: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.232, MCPMod BetaMod model — Adjusted p-value from multiple contrast test; Assumption: 80% of the maximum effect is achieved at the medium dose and the maximum effect is achieved at the 70% of the high dose

2. Secondary Outcome: Part 1 - Percent Change From Baseline in Draining Fistula/Tunnel (dT) Count at Week 16
Description: Percent change from baseline in draining fistula/tunnel (dT) count at Week 16 is reported. Tunnel/fistula/sinus were counted as dT only if draining.
  Least square means and standard errors were estimated by MMRM, which included fixed categorical effects of treatment at each visit, TNFi status at baseline, categorical baseline dT count and fixed continuous effect of baseline of outcome measures at each visit. Visit was treated as repeated measure with an unstructured covariance matrix for the within trial participant variability and all visits with planned measurements of the outcome variable as well as all dose groups were included in the model.
Time Frame: The MMRM model incorporates dT count from baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14 and Week 16. The data represent the Least Squares Means at Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Number analyzed (Participants) | 53 | 53 | 52 | 51
Percentage change | -14.0 (10.6) | -23.5 (10.7) | -36.2 (10.8) | -22.7 (11.2)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab low dose group; The MMRM included fixed categorical effects of treatment at each visit, TNFi status at baseline, categorical baseline dT count and fixed continuous effect of baseline of outcome measures at each visit. Visit was treated as repeated measure with an unstructured covariance matrix for the within trial participant variability and all visits with planned measurements of the outcome variable as well as all dose groups were included in the model; Test type: Other; Difference of least square means = -9.6, 95% CI 2-sided [-39.2 to 20.1], Standard Error of Mean 15.0 — Difference = (least square mean Spesolimab low dose) - (least square mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs Spesolimab medium dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = -22.2, 95% CI 2-sided [-52.0 to 7.6], Standard Error of Mean 15.1 — Difference = (least square mean Spesolimab medium dose) - (least square mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs Spesolimab high dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = -8.8, 95% CI 2-sided [-39.1 to 21.6], Standard Error of Mean 15.4 — Difference = (least square mean Spesolimab high dose) - (least square mean Placebo)

3. Secondary Outcome: Part 1 - Absolute Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) Value at Week 8
Description: IHS4 is a validated, clinical scoring system for dynamic assessment of HS severity. The score was calculated as: (number of nodules x1) + (number of abscesses x2) + (number of draining tunnels [fistulae/sinuses] x4). The minimum is 0, the maximum depends on the count of nodules, abscesses, and draining tunnels. Scores 0-3 indicate mild HS, 4-10 moderate HS, ≥11 severe HS. Absolute change from baseline was calculated as follows: (IHS4 value at visit timepoints) - (IHS4 value at baseline).
  Least square means and standard errors were estimated by MMRM, which included fixed categorical effects of treatment at each visit, TNFi status at baseline, categorical baseline dT count and fixed continuous effect of baseline of outcome measures at each visit. Visit was treated as repeated measure with an unstructured covariance matrix for the within trial participant variability and all visits with planned measurements of the outcome variable as well as all dose groups were included in the model.
Time Frame: The MMRM model incorporates IHS4 value from baseline (Week 0), Week 2, Week 4, Week 6 and Week 8. The data represent the Least Squares Means at Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Number analyzed (Participants) | 53 | 53 | 52 | 51
Units on a scale | -13.5 (2.5) | -11.1 (2.5) | -14.1 (2.5) | -10.5 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab low dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = 2.4, 95% CI 2-sided [-4.5 to 9.4], Standard Error of Mean 3.5 — Difference = (least square mean Spesolimab low dose) - (least square mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs Spesolimab medium dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = -0.6, 95% CI 2-sided [-7.5 to 6.3], Standard Error of Mean 3.5 — Difference = (least square mean Spesolimab medium dose) - (least square mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs Spesolimab high dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = 3.0, 95% CI 2-sided [-3.9 to 10.0], Standard Error of Mean 3.5 — Difference = (least square mean Spesolimab high dose) - (least square mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.887, MCPMod Linear model — Adjusted p-value from multiple contrast test; No assumptions
Statistical Analysis 5: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.902, MCPMod Exponential: model — Adjusted p-value from multiple contrast test; Assumption: 30% of the maximum effect is achieved at the medium dose
Statistical Analysis 6: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.866, MCPMod Emax model — Adjusted p-value from multiple contrast test; Assumption: 70% of the maximum effect is achieved at the medium dose
Statistical Analysis 7: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.825, MCPMod SigEmax model — Adjusted p-value from multiple contrast test; [statistical method as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs Spesolimab low dose group vs Spesolimab medium dose group vs Spesolimab high dose group; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.634, MCPMod BetaMod model — Adjusted p-value from multiple contrast test; [statistical method as in outcome 1, analysis 8]

4. Secondary Outcome: Part 1 - Absolute Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) Value at Week 16
Description: as for outcome 3
Time Frame: The MMRM model incorporates IHS4 from baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14 and Week 16. The data represent the Least Squares Means at Week 16.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Number analyzed (Participants) | 53 | 53 | 52 | 51
Units on a scale | -11.8 (3.8) | -7.2 (3.9) | -17.0 (3.9) | -4.2 (4.0)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab low dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = 4.6, 95% CI 2-sided [-6.1 to 15.3], Standard Error of Mean 5.4 — Difference = (least square mean Spesolimab low dose) - (least square mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs Spesolimab medium dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = -5.2, 95% CI 2-sided [-15.9 to 5.5], Standard Error of Mean 5.4 — Difference = (least square mean Spesolimab medium dose) - (least square mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs Spesolimab high dose group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference of least square means = 7.6, 95% CI 2-sided [-3.3 to 18.5], Standard Error of Mean 5.5 — Difference = (least square mean Spesolimab high dose) - (least square mean Placebo)

5. Secondary Outcome: Part 1 - Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: The occurrence of treatment emergent adverse events (TEAEs) is reported as the number of patients with TEAEs.
Time Frame: From first drug administration until end of exposure, plus residual effect period, up to approximately 68 weeks.
Population: Safety Analysis Set (SAF): all subjects who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
Number analyzed (Participants) | 53 | 53 | 52 | 51
Participants | 44 | 47 | 51 | 47

ADVERSE EVENTS:
Time Frame: From first drug administration until end of exposure (date of last administration - date of first administration +1 day + dosing interval [7 days if last dose was on Week 0-7 or 16-17; 14 days if last dose was on Week 8-14, 18-48]), plus residual effect period, up to approximately 68 weeks.
Description: Safety Analysis Set (SAF): all subjects who were randomized and received at least one dose of study drug.
Groups:
- Spesolimab following placebo: Patients in the placebo group switched from Week 16 until the end of treatment (Week 48) to the same subcutaneous injection (s.c.) dose of spesolimab administered to patients in the medium and high dose groups (starting with 3 loading s.c. doses of spesolimab every week and then maintenance s.c. dose of spesolimab every 2 weeks).
Arm/Group | Placebo | Spesolimab following placebo | Spesolimab low dose group | Spesolimab medium dose group | Spesolimab high dose group
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50 | 0/53 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 3/53 | 7/50 | 3/53 | 8/52 | 6/51
Other Adverse Events (participants affected / at risk) | 29/53 | 32/50 | 39/53 | 38/52 | 41/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Spesolimab following placebo (N=50) | Spesolimab low dose group (N=53) | Spesolimab medium dose group (N=52) | Spesolimab high dose group (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Severe fever with thrombocytopenia syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinoatrial block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Spesolimab following placebo (N=50) | Spesolimab low dose group (N=53) | Spesolimab medium dose group (N=52) | Spesolimab high dose group (N=51)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 4
Nausea (Gastrointestinal disorders) | 4 | 2 | 3 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 3 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 1 | 5
Injection site pain (General disorders) | 3 | 2 | 3 | 2 | 0
Injection site pruritus (General disorders) | 0 | 2 | 2 | 3 | 3
Injection site reaction (General disorders) | 3 | 5 | 5 | 2 | 2
Pyrexia (General disorders) | 3 | 5 | 3 | 0 | 4
Nasopharyngitis (Infections and infestations) | 4 | 0 | 2 | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 9 | 11 | 7
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 9 | 4 | 6 | 6 | 5
Hidradenitis (Skin and subcutaneous tissue disorders) | 9 | 13 | 19 | 10 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 5 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 4
Influenza like illness (General disorders) | 0 | 1 | 3 | 1 | 1
Injection site bruising (General disorders) | 1 | 1 | 1 | 3 | 0
Injection site erythema (General disorders) | 3 | 3 | 1 | 3 | 3
Injection site swelling (General disorders) | 2 | 3 | 0 | 1 | 1
Pain (General disorders) | 4 | 1 | 1 | 2 | 5
COVID-19 (Infections and infestations) | 2 | 4 | 4 | 3 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 3 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 4 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 3 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 2 | 2
Hypertension (Vascular disorders) | 1 | 1 | 3 | 2 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3

LIMITATIONS AND CAVEATS:
The Part 2 was not initiated due to discontinuation of this trial according to protocol. The interim analysis in Part 1 was done after all patients reached Week 16 milestone, and following the analysis, the decision to discontinue was taken.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT05819398/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT05819398/SAP_001.pdf